CLINICAL TRIAL: NCT06389227
Title: Developing the Physical Performance in Youth Soccer: Short-term Effect of Dynamic-Ecological Versus Traditional Training Approach for Sub-élite U13 Players: An Ecological Exploratory Cluster Randomised Trial
Brief Title: Developing the Physical Performance in Youth Soccer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0433611
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Motor Activity
Keywords: ecological dynamic approach; motor performance ability; soccer performance; young soccer player
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dynamic-ecological approach (DEA) (Experimental): The DEA completed 18 ninety-minute sessions (3 per week) for six weeks oriented to soccer training using the dynamic ecological approach
  Interventions: Other: dynamic ecological approach (DEA)
- traditional training group (TTG) (Active Comparator): TTG followed a traditional soccer training program for the same period and number of ses-sions without any intervention attributable to the dynamic ecological approach
  Interventions: Other: traditional training group

INTERVENTIONS:
Other: dynamic ecological approach (DEA) — The DEA completed 18 ninety-minute sessions (3 per week) for six weeks oriented to soccer training using the dynamic ecological approach
  Arms: dynamic-ecological approach (DEA)
Other: traditional training group — The TTG followed a traditional soccer training program for the same period and number of sessions without any intervention attributable to the dynamic ecological approach
  Arms: traditional training group (TTG)

SUMMARY:
Therefore, this study aims to verify the effects of a soccer training program based on the dynamic-ecological approach on U13 sub-elité players' physical efficiency by analysing explosive strength, speed, resistance to speed and muscle flexibility. This study hypothe-sises that the dynamic-ecological approach can consistently help players develop adequate physical efficiency and motor coordination.

DETAILED DESCRIPTION:
Nowadays, research in youth soccer consists of methodological choices that can raise ac-tivity volumes and exercise intensity to promote proper training for youth soccer de-mands. Therefore, the present cluster randomised trial aims to evaluate the effects on physical performance parameters of the dynamic-ecological approach compared with a traditional one in a group of sub-élite U13 players. Thirty-five male children (age 12.16 ± 0.55 years; weight 45.59 ± 7.15 kg; height 145.5 ± 4.2 cm; BMI 15.8 ± 2.1 kg*m-²) were re-cruited for this trial from two teams belonging to sub-élite soccer schools and randomly assigned in a dynamic-ecological approach (DEA) or a traditional training (TTG) group. The training program lasted six weeks and consisted of 18 training sessions of 90 minutes each (3 sessions per week). The sample was evaluated by Standing Long Jump (SLJ), hop test (HT), 10 m sprint (10m), 10 x 5 m shuttle run test (SRT) and Leg Raise test (LR). The DEA group showed significantly higher results in the SLJ (p< .001), HT left leg (p<.001), 10m sprint (p<.001), and SRT (p<.001). In conclusion, the dynamic-ecological approach provides higher performance adaptations. Therefore, this approach can be considered a suitable method to optimise prepubertal player training, mainly when no fitness or strength coach is available.

ELIGIBILITY:
Inclusion Criteria:

* had not suffered an injury in the previous 6 months;
* who, in the 4 weeks before the study, had systematically performed the training sessions without interruptions or absences;
* all those who, upon medical evaluation, fell within stages 3 and 4 of Tanner's classification

Exclusion Criteria:

-Goalkeepers and players who had been injured in the previous six months or did not meet the established minimum compliance were excluded from this study

Ages: 12 Years to 13 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Thirty-five male children under 13 years old
Enrollment: 35 (Actual)
Dates: Start 2023-10-15 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Number of participants evaluated on physical efficiency | From enrollment to the end of the study at six weeks
  Direct outcome measurements pre-test vs post-test, Intervention vs treatment

CONTACTS AND LOCATIONS:
Overall Officials: Federico Abate Daga, MSC PhD, Principal Investigator — University of Turin, Italy
Locations (1):
- Cit Turin LDE, Turin, Italy

IPD SHARING:
Plan to Share IPD: No
Italian GDPR law